CLINICAL TRIAL: NCT06730607
Title: Image-Based Prediction of Ventricular Tachycardia Events in Post-Myocarditis Patients: an International Multicenter Case-control Study
Brief Title: Image-Based Prediction of Ventricular Tachycardias in Post-Myocarditis Patients: an International Multicenter Case-control Study
Acronym: MYOCARDITIS-VT
Status: Recruiting | Type: Observational
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of Arrhythmia Department, Centro Medico Teknon
Other Study IDs: MYOCARDITIS-VT
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Myocarditis; Ventricular Arrhythmia
Keywords: myocarditis; ventricular arrhythmias; sudden cardiac death; cardiac magnetic resonance
MeSH Terms: conditions — Myocarditis; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: patients with sudden cardiac death or sustained ventricular arrhythmias during the follow-up: Inclusion criteria
  Patients will only be recruited if they fulfill ALL the inclusion criteria:
  1. Age > 18 years.
  2. Myocarditis diagnosis > 6 months before the inclusion in the study.
  3. Signed informed consent.
  4. CMR performed > 6 months after myocarditis diagnosis
  Exclusion criteria
  Patients will be excluded if they meet ANY of the following exclusion criteria:
  * Age < 18 years.
  * Pregnancy.
  * Other concomitant structural heart diseases (e.g. congenital, non-ischemic, etc.)
  * Active myocarditis
  * Myocarditis diagnosis < 6 months
  * Previously documented sustained ventricular arrhythmias.
  * Impossibility or contraindications to undergo LGE-CMR.
  * Concomitant investigation treatments.
  * Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.
- Controls:patients without sudden cardiac death or sustained ventricular arrhythmias during follow-up: Patients will only be recruited if they fulfill ALL the inclusion criteria:
  1. Age > 18 years.
  2. Myocarditis diagnosis > 6 months before the inclusion in the study.
  3. Signed informed consent.
  4. CMR performed > 6 months after myocarditis diagnosis
  Patients will be excluded if they meet ANY of the following exclusion criteria:
  * Age < 18 years.
  * Pregnancy.
  * Other concomitant structural heart diseases (e.g. congenital, non-ischemic, etc.)
  * Active myocarditis
  * Myocarditis diagnosis < 6 months
  * Previously documented sustained ventricular arrhythmias.
  * Impossibility or contraindications to undergo LGE-CMR.
  * Concomitant investigation treatments.
  * Medical, geographical and social factors that make study participation impractical, and

SUMMARY:
Ventricular arrhythmias (VAs) are frequently associated with structural heart diseases (SHD) such as myocardial infarction, myocarditis, and non-ischemic cardiomyopathies. Myocardial fibrotic tissue plays a central role in the genesis and the maintenance of re-entrant VAs associated with post-myocarditis sequelae and late gadolinium enhancement cardiac magnetic resonance (LGE-CMR) has proven to be a useful tool for the non-invasive characterization of the scarred tissue and the underlying arrhythmogenic substrate. Moreover, a post-processing imaging platform named ADAS 3D LV (ADAS3D Medical SL, Barcelona, Spain) allows to analyze the CMR-derived data and to characterize the scar architecture, differentiating between dense (scar core zone) and more diffuse (border zone [BZ]) fibrosis, and identifying the BZ channels (BZCs) that are strands of healthy myocardial tissue within zones of unexcitable tissue and connect areas of normal myocardium. It was described that BZCs could serve as slow-conducting reentrant pathways and are critical to entail VA in ischemic and non-ischemic heart disease. However, the pathophysiological role and the correlation between scar architecture and VAs in post-myocarditis patients is yet to be defined.

To date, the standard-of-care evaluation for primary prevention implantable cardioverter-defibrillator (ICD) therapy is LVEF-based, leading to the fact that the contemporary rate of appropriated therapies is very low. Moreover, events may also occur in patients with normal to moderately depressed LVEF, which is particularly relevant, as it constitutes the most prevalent population of patients exposed to an increased risk of VAs. Multiple studies reported that LGE at CMR is a strong and specific predictor of VT occurrence and sudden death in post-myocarditis patients. There were reported cases in which even after the normalization of LVEF, the extension of LGE, the scar architecture, and the presence of BZCs at cMR analysis are determinants of the arrhythmic risk in post-myocarditis patients.

The Investigators sought to evaluate the usefulness of CMR-derived scar architecture analysis to predict the occurrence of VT events in an international, multicenter, case-control study on unselected post-myocarditis patients without previous arrhythmia evidence. Aim of the study is also to assess the net reclassification improvement (NRI) for the indication of primary prevention ICD implantation using CMR data and post-processing data as compared to LVEF-based indication

DETAILED DESCRIPTION:
Research hypothesis

The composite outcome is:

* sudden cardiac death, sustained VT, syncopal VT or appropriate ICD therapy (ATP and/or shock) in ICD carriers in primary prevention, or
* sudden cardiac death, sustained VT, syncopal VT detected by any diagnostic test (i.e., 24 h Holter monitoring, prolonged Holter monitoring, urgency ECG etc.) in no ICD-carriers.

Our research hypothesis is that the composite outcome will be higher in those patients with greater scar mass and BZC mass.

Primary objective To analyze the composite outcome of sudden cardiac death or sustained ventricular tachycardia (either treated by an ICD or documented by any diagnostic method) in post-myocarditis patients with no previous arrhythmia evidence, according to their risk classification by means of BZC mass.

Secondary objectives

To analyze the relationship between the primary outcome and other variables:

* LVEF
* Scar mass
* BZ mass
* Core mass
* Presence and number of tissue channels within the scar, as detected by cardiac CT
* Age
* Time since myocarditis

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Myocarditis diagnosis > 6 months before the inclusion in the study.
3. Signed informed consent.
4. CMR performed > 6 months after myocarditis diagnosis

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Other concomitant structural heart diseases (e.g. congenital, non-ischemic, etc.)
* Active myocarditis
* Myocarditis diagnosis < 6 months
* Previously documented sustained ventricular arrhythmias.
* Impossibility or contraindications to undergo LGE-CMR.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previous myocarditis and a cardiac magnetic resonance performed at least 6 months after the diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients presenting one of sudden cardiac death, sustained ventricular arrhythmia, or defibrillator therapy. | 2 years
  The primary endpoint will be the clinical composite of sudden cardiac death or any sustained ventricular arrhythmia.
  The endpoint will be retrospectively correlated with the cMR-derived findings.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Humanitas Research Hospital, Rozzano, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, Pisa
- Teknon Medical Center, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acosta J, Fernandez-Armenta J, Borras R, Anguera I, Bisbal F, Marti-Almor J, Tolosana JM, Penela D, Andreu D, Soto-Iglesias D, Evertz R, Matiello M, Alonso C, Villuendas R, de Caralt TM, Perea RJ, Ortiz JT, Bosch X, Serra L, Planes X, Greiser A, Ekinci O, Lasalvia L, Mont L, Berruezo A. Scar Characterization to Predict Life-Threatening Arrhythmic Events and Sudden Cardiac Death in Patients With Cardiac Resynchronization Therapy: The GAUDI-CRT Study. JACC Cardiovasc Imaging. 2018 Apr;11(4):561-572. doi: 10.1016/j.jcmg.2017.04.021. Epub 2017 Aug 2. PMID 28780194
- [Background] Jauregui B, Soto-Iglesias D, Penela D, Acosta J, Fernandez-Armenta J, Linhart M, Ordonez A, San Antonio R, Teres C, Chauca A, Carreno JM, Scherer C, Falasconi G, Prat-Gonzalez S, Perea RJ, Mont L, Bosch X, Ortiz-Perez JT, Berruezo A. Cardiovascular magnetic resonance determinants of ventricular arrhythmic events after myocardial infarction. Europace. 2022 Jul 15;24(6):938-947. doi: 10.1093/europace/euab275. PMID 34849726
- [Background] Di Marco A, Brown P, Mateus G, Faga V, Nucifora G, Claver E, Viedma J, Galvan F, Bradley J, Dallaglio PD, de Frutos F, Miller CA, Comin-Colet J, Anguera I, Schmitt M. Late gadolinium enhancement and the risk of ventricular arrhythmias and sudden death in NYHA class I patients with non-ischaemic cardiomyopathy. Eur J Heart Fail. 2023 May;25(5):740-750. doi: 10.1002/ejhf.2793. Epub 2023 Feb 22. PMID 36781200
- [Background] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965